CLINICAL TRIAL: NCT05753878
Title: A Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetic and Immunogenicity of HH-120 Nasal Spray in Healthy Subjects
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of HH-120 Nasal Spray in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Huahui Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HH120-NS111
Record Dates: First submitted 2023-02-23; First posted 2023-03-03 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- HH-120 nasal spray, Part A cohort 1 (Experimental): Nasal endoscopic examination is performed at 3min (±2 min), 30min (±5 min), 1h (±10 min), and 2h (±10 min) after dosing.
  Interventions: Drug: HH-120 nasal spray, PartA cohort 1
- HH-120 nasal spray, Part A cohort 2-7 (Experimental): Nasal/nasopharyngeal samples are collected at 3min (±2 min) , 1h (±10 min) ,2h (±10 min),4h (±30 min),8h (±30 min),24h (±30 min).
  Interventions: Drug: HH-120 nasal spray, Part A cohort 2-7
- HH-120 nasal spray, Part A cohort 8-9 (Experimental): Nasal/nasopharyngeal samples are collected at 4h (±30 min) , 8h (±30 min).
  Interventions: Drug: HH-120 nasal spray, Part A cohort 8-9
- HH-120 nasal spray, Part B (Experimental)
  Interventions: Drug: HH-120 nasal spray, Part B
- Placebo nasal spray, Part B (Placebo Comparator)
  Interventions: Other: Placebo nasal spray, Part B

INTERVENTIONS:
Drug: HH-120 nasal spray, PartA cohort 1 — A single dose of HH-120 nasal spray premixed with 1mg/ml methylene blue injection.
  Arms: HH-120 nasal spray, Part A cohort 1
Drug: HH-120 nasal spray, Part A cohort 2-7 — A single dose of HH-120 nasal spray.
  Arms: HH-120 nasal spray, Part A cohort 2-7
Drug: HH-120 nasal spray, Part A cohort 8-9 — Two doses of HH-120 nasal spray.
  Arms: HH-120 nasal spray, Part A cohort 8-9
Drug: HH-120 nasal spray, Part B — HH-120 nasal spray, 10 times daily for 7 consecutive days.
  Arms: HH-120 nasal spray, Part B
Other: Placebo nasal spray, Part B — Placebo nasal spray, 10 times daily for 7 consecutive days.
  Arms: Placebo nasal spray, Part B

SUMMARY:
This is a clinical study evaluating the safety, tolerability, pharmacokinetic (PK) characteristics and immunogenicity of HH-120 nasal spray in healthy subjects. This study is divided into two parts: Part A is of open-label design and mainly aims to assess the local distribution and PK in nasal cavity of HH-120 nasal spray, subjects from 10 cohorts are sequentially enrolled to perform either nasal endoscopic examination or nasal/ nasopharyngeal samples collection at different time points post administration. Part B mainly aims to assess the safety, systematic pharmacokinetic and immunogenicity after multiple dosing of HH-120 nasal spray, subjects are randomly assigned (3:1) to HH-120 and placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 to 65 (including 18 and 65 years old);
* The weight of male subjects is not less than 50 kg, and the weight of female subjects is not less than 45 kg. Body Mass Index (BMI) = weight (kg)/height2 (m2), BMI is within the range of 18~28kg/m2 (including the critical value);
* Normal physical examination, vital signs, laboratory tests and other auxiliary examinations (chest imaging, abdominal B-ultrasound, electrocardiogram, etc.) or abnormality without clinical significance.
* Willing and able to give written informed consent.

Exclusion Criteria:

* Participated in any other clinical research with drug intervention within 4 weeks before screening, or the drug is still in the elimination period (5 half-lives) before screening, whichever is longer;
* Have used therapeutic biological agents within 12 weeks before screening, or are within the drug elimination period (5 half-lives) at the time of random administration, whichever is longer;
* Have been vaccinated within 12 weeks before screening, or plan to receive BCG or other vaccines during the study or within 12 weeks after the study;
* Have used any prescription drugs, non-prescription Chinese herbal medicines or health products within 14 days (inclusive) before the screening;
* Have undergone any major surgery within 8 weeks (including 8 weeks) before screening, or need to undergo such surgery during the study period, and deemed by the investigator and the sponsor that such surgery may bring unacceptable risk to the subject.;Physical examination, laboratory abnormalities, and medical history;
* Supine systolic blood pressure (SBP) >140mmHg or <90 mmHg, and/or diastolic blood pressure (DBP) >90mmHg or <50 mmHg during the screening period;
* Supine 12-lead electrocardiogram showing QTcF interval > 450 ms (male) or > 470 ms (female). and/or other abnormalities with clinical significance during screening;
* History of systemic or respiratory infection within 2 weeks before screening, or concurrent viral or bacterial infection (fever or other symptoms) during screening;
* Have received vital organ transplantation (such as heart, lung, liver, kidney, etc.);
* Have malignant tumor diseases (excluding malignant tumors that have been cured and have no recurrence within the past 5 years, completely resected basal cell and squamous cell skin cancers, and completely resected carcinoma in situ of any type);
* Hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (Anti-HCV), Treponema pallidum antibody and acquired immunodeficiency syndrome (HIV) antibody positive;
* History of cardiovascular system, digestive system, kidney, liver, endocrine system, blood and lymphatic system, immune, nervous system or mental disorders or any other significant diseases, or suffer from chronic rhinitis or allergic rhinitis, drug abuse, alcoholism
* Have a history of drug abuse or used drugs in the past six months or have a positive urine drug screening;
* Have a history of alcoholism or excessive alcohol intake in the past 6 months (drinking 14 units of alcohol per week: 1 unit = 285mL of beer, or 25mL of spirits, or 100mL of wine), or those who have a positive alcohol breath test; or test Cannot cooperate with non-drinkers during the period;
* Known hypersensitivity to any ingredient used in the dosage form of intervention therapy; ever hypersensitivity (regardless of degree) to other monoclonal antibody drugs and therapeutic protein preparations (fresh or frozen plasma, human serum albumin, cytokines, interleukins, etc.) ; or have a clear past allergy to inhalant allergens (regardless of degree);
* History of severe allergic reactions or hypersensitivity reactions, or those with allergic constitution (allergic to multiple drugs and food);
* Have child-bearing plan or are unable to voluntarily take effective contraceptive measures, or plan to donate sperm/ovum;
* Positive for human chorionic gonadotropin (β-Human Chorionic Gonadotropin, β-HCG) or are breastfeeding;
* Have blood losing >400mL in the past 3 months, or have received blood transfusion; or plan to donate blood during the study;
* Any other circumstances that the researchers deemed not suitable for participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
The distribution of HH-120 in the nasal cavity at different time points after single dose of HH-120 nasal spray.(Part A: cohort 1) | From baseline to the end of the 7-day follow-up.
Local drug concentration of nasal and nasopharyngeal swab samples before and at different time points after dosing of HH-120 nasal spray.(Part A: cohort 2-9) | From baseline to the end of the 7-day follow-up.
The incidence and severity of adverse events and the serious adverse events.(Part B) | From baseline to the end of the 29-day follow-up.

SECONDARY OUTCOMES:
The incidence and severity of adverse events and the serious adverse events.(Part A) | From baseline to the end of the 7-day follow-up.
Drug concentration of nasopharyngeal swab samples before and after multiple dosing of HH-120 nasal spray.(Part B) | From baseline to the end of the 29-day follow-up.
Maximum plasma concentration (Cmax).(Part B) | From baseline to the end of the 29-day follow-up.
Peak time (Tmax).(Part B) | From baseline to the end of the 29-day follow-up.
The incidence and titer of anti-drug antibody (ADA).(Part B) | From baseline to the end of the 29-day follow-up.

OTHER OUTCOMES:
The in vitro SARS-CoV-2 neutralization activity of nasal and nasopharyngeal swab samples at different time points after dosing.(Part A) | From baseline to the end of the 7 days follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing TongRen Hospital, Capital Medical University, Beijing, Beijing Municipality, China